CLINICAL TRIAL: NCT00645268
Title: A Multicenter, Double-blind Study to Evaluate the Effect of Pretreatment With a Daily Dose of Viagra® (Sildenafil Citrate) on the PRN Efficacy of Viagra in Men With Erectile Dysfunction and Type 2 Diabetes
Brief Title: A Multicenter, Double-blind Study to Evaluate the Effect of Pretreatment With a Daily Dose of Sildenafil on the As-Needed Efficacy of Viagra in Men With Erectile Dysfunction and Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481146
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Erectile Dysfunction; Diabetes Mellitus, Type 2 | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 2 (Placebo Comparator)
  Interventions: Drug: placebo
- Open-Label Arm (Other)
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — In the double-blind phase, patients received sildenafil 50 mg once daily during Week 1 (7 doses), followed by a daily dose of sildenafil 100 mg during the next 3 weeks.
  Arms: Arm 1
Drug: placebo — In the double-blind phase, patients received placebo once daily during Week 1 (7 doses), followed by a daily dose of placebo during the next 3 weeks.
  Arms: Arm 2
Drug: sildenafil — Eligible subjects then entered an open-label phase during which all subjects received sildenafil 50 mg as needed for sexual activity for the next 2 weeks, which could be titrated to either 25 mg or 100 mg based on the investigator's assessment of efficacy and tolerability, for 10 weeks (12 weeks total).
  Arms: Open-Label Arm

SUMMARY:
To determine the effect on erectile function in a population of type 2 diabetic men with erectile dysfunction who have undergone the following treatment regimen: pre-treatment with a daily dose of double-blind sildenafil versus placebo for 4 weeks (Phase I) followed by an as-needed, flexible-dose, open-label treatment phase with sildenafil for 12 weeks (Phase II). To assess safety and tolerability of this dosing regimen and to investigate its effects on endothelial function and subject's responses to the Self-Esteem And Relationship (SEAR) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Patients had a documented clinical diagnosis of erectile dysfunction, a sexual partner for the duration of the study, and have a HbAlc of less than or equal to 10 at screening. Type 2 diabetic patients currently on insulin or on combination therapy with an oral hypoglycemic agent were not excluded.

Exclusion Criteria:

Excluded were subjects who had taken more than 6 doses of any PDE5 inhibitor and/or had taken their last dose less than 4 weeks prior to the screening visit; subjects with resting sitting and/or standing hypotension (BP < 90/50mmHg) or hypertension (BP > 170/110mmHg); and subjects with significant cardiovascular disease, including cardiac failure, myocardial infarction, unstable angina, stroke or transient ischemic attack (TIA), symptomatic or clinically significant cardiac arrhythmias including atrial fibrillation in the last 3 months.

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2002-12; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
The IIEF Erectile Function (EF) Domain score | Week 4

SECONDARY OUTCOMES:
Intercourse success rate based on Event Logs | continuous
Ability to obtain an erection hard enough to attempt sexual intercourse post dose of sildenafil | continuous
Responses to the Self-Esteem And Relationship (SEAR) Questionnaire (including individual domain scores for the Sexual Activity, Self-Esteem And Relationship domains) | Week 16
Responses to International Index of Erectile Function (IIEF) and secondary IIEF Domain scores (Orgasm; Desire; Intercourse Satisfaction; Overall Satisfaction) | Week 16
Reponses to the Global Efficacy Assessment Questions | Week 16
Flow mediated brachial artery dilation (FMD) as an index of generalized endothelial function | Week 4, 6, and 16

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (24):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Laguna Woods, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, New Albany, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Richmond Heights, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Pfizer Investigational Site, Calgary, Canada

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481146&StudyName=A%20Multicenter%2C%20Double-blind%20Study%20to%20Evaluate%20the%20Effect%20of%20Pretreatment%20With%20a%20Daily%20Dose%20of%20sildenafil%20on%20the%20As-Needed%20Efficacy%20o